CLINICAL TRIAL: NCT05150327
Title: Multicenter Retrospective Cohort Study of Invasive Fungal Filamentous Fungal Infections in Liver Transplant Patients
Brief Title: Multicenter Cohort Study of Invasive Fungal Filamentous Fungal Infections in Liver Transplant Patients
Acronym: FongiFoie
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8429
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fungal Infection
Keywords: Fungal Infection; Immunodeficiency; Fungal filamentous; Liver transplant; Organ transplant
MeSH Terms: conditions — Mycoses; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Invasive filamentous fungal infections (aspergillosis, scedosporiosis, mucormycosis, fusarium wilt) are frequent and serious in immunocompromised individuals and especially in organ transplant patients. There is little recent data in liver transplantation, especially on the incidence and risk factors of fungal infections

ELIGIBILITY:
Inclusion Criteria

* Age: from birth
* Subject with a liver transplant in one of the centers participating in the study
* Invasive fungal infection with filamentous fungus between 2007-2021
* Proven or probable infection with filamentous fungi according to EORTC/MSGERC criteria:

  * Invasive aspergillosis
  * Mucormycosis
  * Fusariosis
  * Scedosporiosis
  * Other infection with filamentous fungus
* Subject or legal representative for minors, who has not expressed, after information, his opposition to the reuse of his data for scientific research purposes.

Exclusion Criteria

* Subject or (legal representative for minors) who has expressed his opposition to participating in the study
* Subject not with a liver transplant
* Subject under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with liver transplantation with proven nvasive fungal infection with filamentous fungus between 2007-2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Study of the incidence, risk factors and prognostic factors associated with invasive fungal filamentous fungal infections in liver transplant patients. | Files analysed retrospectively from January 01, 2007 to December 31, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: François DANION, MD, Study Director — Service des Maladies Infectieuses et Tropicales - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service des Maladies Infectieuses et Tropicales - Hôpitaux Universitaires de Strasbourg, Strasbourg, France